CLINICAL TRIAL: NCT00808171
Title: Evaluation of the Analgesy Using a Local Anesthetic (Lidocaine and Prolocaine) Eutectic Mixture and/or Nitric Oxide at 50% in Oxygen (Livopan®) in Pediatric Patients That During Lumbar Puncture
Brief Title: Evaluation of the Analgesy With Emla and/or Nitrous Oxide in Pediatric Patients for Lumbar Puncture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Renato Santiago Gomez, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CAAE0450020300008
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia; Non Hodgkin Lymphoma
Keywords: lumbar punction; myelogram; pain assessment; nitrous oxide and EMLA; Leukemia and non Hodgkin lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin | interventions — Oxygen; Prilocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EMLA and Livopan (Experimental): Administered EMLA and Livopan
  Interventions: Drug: Livopan; Drug: EMLA
- EMLA and gas placebo (Experimental): Administered EMLA and oxygen
  Interventions: Drug: EMLA
- Livopan and placebo cream (Experimental): Administered Livopan and placebo cream
  Interventions: Drug: Livopan

INTERVENTIONS:
Drug: Livopan — Inhalation of oxygen and nitrous oxide 50%
  Other Names: equimolar mixture of nitrous oxide/oxygen
  Arms: EMLA and Livopan
Drug: Livopan — equimolar mixture of N2O/O2
  Other Names: equimolar mixture of nitrous oxide/oxygen
  Arms: Livopan and placebo cream
Drug: EMLA — Lidocaine-prilocain cream
  Other Names: Eutetic mixture of local anesthetics lidocaine/prilocaine
  Arms: EMLA and Livopan; EMLA and gas placebo

SUMMARY:
In this randomised controlled study the investigators intended to compare the analgesic effects of EMLA and\or nitrous oxide in children submitted to lumbar puncture.

DETAILED DESCRIPTION:
It is a randomized controlled clinical trial, double blinded, with the purpose to compare the use of EMLA - local anesthetic (lidocaine and prilocaine), and or nitrous oxide at 50% in oxygen (Livopan®) to prevent and treat pain in pediatric patients aged four to 16 years old submitted to lumbar puncture for intrathecal chemotherapy. Pain was assessed using the Wong Baker faces scale and the visual numeric scale during six observational periods: baseline; three minutes after gas administration and before the first attempt of lumbar puncture; during the first lumbar puncture attempt; during the chemotherapy administration; during needle remove and three minutes after gas interruption. All the studied procedures will have clinical indication and will not be held by the researcher. The children was random divided within three groups A, B and C as follow: Group A (n=16)EMLA + Livopan; Group B (n=19)EMLA + gas placebo (oxygen); Group C (n=17) Livopan® + placebo cream.

Primary outcome was the detection of a difference of 20% or more in the visual numeric scale between the three treatment groups during the first attempt of lumbar puncture.

ELIGIBILITY:
Inclusion Criteria:

* Age between four and 14 years;
* Not present cognitive disabilities;
* Necessity to perform the clinical procedure;
* Accordance in participating in the study.

Exclusion Criteria:

* Continuity skin lesion in the procedure site;
* Metahemoglobinemia;
* Neuromuscular disability;
* Presence of pneumothorax, emphysema, intra-abdominal infection, cranioencephalic traumatism, otitis media, sinusitis and intracranial hypertension;
* Vitamin B12 known deficits;
* Urgency for the procedure;
* Disagreement in participating of the project;
* Patients in use of Dapsone.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2009-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Compare analgesic efficacy of EMLA versus Nitrous oxide | Within first hour after the procedures

SECONDARY OUTCOMES:
Evaluate analgesic synergism of EMLA versus nitrous oxide | One hour after the procedures

CONTACTS AND LOCATIONS:
Overall Officials: Yerkes P Silva, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Department of Pediatrics - Hematology section - Clinical Hospital of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Steedman B, Watson J, Ali S, Shields ML, Patmore RD, Allsup DJ. Inhaled nitrous oxide (Entonox) as a short acting sedative during bone marrow examination. Clin Lab Haematol. 2006 Oct;28(5):321-4. doi: 10.1111/j.1365-2257.2006.00807.x. PMID 16999723